CLINICAL TRIAL: NCT00841126
Title: An Open, Randomized, Controlled, Parallel Group, Phase III Study to Investigate the Safety and Efficacy of Fermagate and Lanthanum Carbonate Together With a Randomized Placebo Controlled Double Blind Fermagate Comparison in Hemodialysis Patients With Hyperphosphatemia
Brief Title: Phase III Study to Investigate the Safety and Efficacy of Fermagate and Lanthanum Carbonate
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ineos Healthcare Limited (Industry)
Responsible Party: Chief Medical Officer, INEOS Healthcare Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT 401; 2008-004729-41 (EudraCT Number)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Kidney Failure
Keywords: Hyperphosphatemia; Phosphate binder
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — iron-magnesium hydroxycarbonate; lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Magnesium iron hydroxycarbonate (Experimental)
  Interventions: Drug: Magnesium iron hydroxycarbonate
- Lanthanum carbonate (Active Comparator)
  Interventions: Drug: Lanthanum carbonate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium iron hydroxycarbonate — 500 mg tablets, administered orally: initial dosage 500 or 1000 mg (total daily dose 1500 or 3000 mg) depending on serum phosphate concentration, titrated to a maximum DAILY dose of 9000 mg). The total daily dose should be divided and taken with meals. Any SINGLE dose should not exceed 3000 mg.
  Other Names: Alpharen, magnesium iron hydroxycarbonate
  Arms: Magnesium iron hydroxycarbonate
Drug: Lanthanum carbonate — 750 mg chewable tablets, administered orally: initial dosage 750 mg up to 3-times daily (total daily dose 2250 mg), titrated to a maximum SINGLE dose of 1500 mg (DAILY dose 3750 mg). The total daily dose should be divided and taken with meals.
  Other Names: Fosrenol
  Arms: Lanthanum carbonate
Drug: Placebo — 0 mg (500 mg-size) tablets, administered orally: The total daily dose should be divided and taken with meals. Any SINGLE dose should not exceed 6 tablets.
  Arms: Placebo

SUMMARY:
Magnesium iron hydroxycarbonate is a phosphate binder that absorbs phosphate from food, reducing the amount that the body can absorb.

The purpose of this study is to assess the efficacy of magnesium iron hydroxycarbonate in subjects requiring hemodialysis, compared with a marketed phosphate binder, lanthanum carbonate and placebo.

DETAILED DESCRIPTION:
High levels of phosphate in the blood are linked with serious effects, due to calcium imbalances (high levels of parathyroid hormone (PTH), bone disease, formation of calcium deposites in the body and blood-vessel disease.

Current guidelines indicate that blood phosphorous levels should be maintained between 1.13 to 1.78 mmol/L in patients who receive hemodialysis.

This is a 2-stage re-randomization design where Stage 1 is a randomized, open label comparison between fermagate and lanthanum carbonate (in a non-inferiority design) and Stage 2 is a randomized double blind comparison between fermagate and placebo (in a superiority design).

Objectives at Stage 1:

Primary Objective:

The primary objective is to establish the efficacy of fermagate by demonstrating the noninferiority (with possible assessment of superiority) of fermagate to lanthanum carbonate in lowering serum phosphate in hemodialysis patients.

Secondary objectives:

The secondary objectives are to:

1. Determine the safety of fermagate in hemodialysis patients.
2. Compare the effects of fermagate and lanthanum carbonate on measures of mineral metabolism, albumin, pre-albumin and iron status.

Objectives at Stage 2:

Stage 2 will use patients who complete the 3-month maintenance period of Stage 1 and who were originally randomized to fermagate.

Primary Objective:

The primary objective is to establish efficacy of fermagate by demonstrating the superiority of fermagate over placebo in lowering serum phosphate in hemodialysis patients.

Secondary objectives:

The secondary objectives are to:

1. Determine the safety of fermagate in hemodialysis patients.
2. Compare the effects of fermagate and placebo on measures of mineral metabolism, albumin, pre-albumin and iron status.

ELIGIBILITY:
Inclusion:

Subjects will be considered eligible for entry in the study if they meet all of the following criteria.

1. Male or female, aged ≥18 years.
2. Able to comply with the study procedures and medication.
3. Written informed consent given.
4. On a stable hemodialysis regimen (at least 3x per week) for ≥12 weeks prior to screening.
5. (a) Subject receiving phosphate binder medication(s) at screening, must have been on a stable regimen (dose and medication) for at least 1 month prior to screening and will remain on this regimen until entry into the washout period OR(b) Subjects (i) is not currently receiving any phosphate binding medication at screening (or medication likely to act as a phosphate binder) and (ii) must not have done so for at least one month and (iii) has sustained hyperphosphatemia.
6. Willing to abstain from taking any phosphate binder or oral magnesium-, oral aluminum- or oral iron-containing products and preparations other than the study medication.
7. If required to take >6000 mg/day of fermagate, the subject will be willing to have at least three meals per day.

   Specifically, for randomization and inclusion into the treatment period, one of the following criteria must be fulfilled:
8. (a) Is not receiving phosphate binding medication at screen and has a screen serum phosphate value above 3.0 mmol/L (9.3 mg/dL)OR(b) Has a serum phosphate value of ≥1.94 mmol/L (≥6.0 mg/dL) at Washout Visit 2 to 4 or above 3.0 mmol/L (9.3 mg/dL) at visit 1 during washout.

Exclusion:

Subjects will not be considered eligible for entry in the study if they meet one or more of the following criteria.

1. Participation in any clinical trial using an investigational product or device during the 30 days preceding the Screening Visit.
2. Previous experience of fermagate treatment.
3. A significant history of alcohol, drug or solvent abuse in the opinion of the investigator.
4. Any disease or condition, physical or psychological that, in the opinion of the investigator, would compromise the safety of the subject or the likelihood of achieving reliable results or increase the likelihood of the subject being withdrawn.
5. Laboratory findings at screening which, in the opinion of the investigator, are clinically significant for this subject population.
6. A screen serum magnesium concentration of >3.0 mg/dL (>1.25 mmol/L).
7. A known history of hemochromatosis.
8. Subjects receiving either tetracycline or lithium treatment.
9. Subjects receiving nicotinamide (niacinamide) or niacin (nicotinic acid) alone (i.e. not as a constituent of a multivitamin supplementation).
10. A serum ferritin level of ≥1500 ng/mL (≥3370 pmol/L).
11. Non-elective hospitalization in the 4 weeks prior to screening.
12. Female subjects who are of childbearing potential and who are neither surgically sterilized nor using reliable contraceptive methods (hormonal, barrier methods or intrauterine device) or who are lactating or pregnant.
13. Current hypophosphatemia at screening (last 2 consecutive phosphate values of <2.2 mg/dL [<0.7 mmol/L]).
14. Known history of colorectal malignancy, familial polyposis coli and/or strong family history (in 2 or more first degree relatives) of these terms
15. A QTcF interval of >560 ms at screen.
16. Known persistent (>1 month) non compliance (<70%) with prescribed medication regimens at screen.
17. Current clinically significant intestinal motility disorder.
18. Intestinal motility disorder with current or previous use of lanthanum carbonate.
19. Known intolerance to lanthanum carbonate or any excipients of fermagate or Fosrenol medication.
20. Subjects with inflammatory bowel disease that, in the investigator's opinion, is poorly controlled.
21. Subjects placed under guardianship or tutelage.
22. Subjects previously withdrawn from the study.

The above inclusion and exclusion criteria would be the same for all countries except the exclusion criteria of the QTc interval would be different for Germany (QTc interval of >470ms at screen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Control or not the level of serum phosphate | Within the treatment period
Stage 2: Change from treated baseline in mean serum phosphate | At 4 weeks

SECONDARY OUTCOMES:
Stage 1: Change from baseline in mean serum phosphate | End of 3 months treatment in maintenance period
Stage 1: Change from baseline in calcium, calcium phosphate product and PTH level | End of 3 months treatment in maintenance period
Stage 2: Change from treated baseline in mean serum phosphate | At weeks 1, 2 and 3
Stage 2: Change from treated baseline in Ca, Ca-phosphate product and PTH levels | At the end of weeks 1, 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Information at Ineos Healthcare Limited (Chief Medical Officer), Study Chair — INEOS Healthcare Ltd, UK
Locations (111):
- United States (62):
  - Nephrology Associates PC, Birmingham, Alabama
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - Southwest Kidney Institute, Tempe, Arizona
  - US Renal Care, Jonesboro, Arkansas
  - Wright Steven (Private Practice), Pine Bluff, Arkansas
  - University of Southern California, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - North America Research Institute, San Dimas, California
  - Kidney Center Inc., Simi Valley, California
  - Nephrology Educational Services and Research, Tarzana, California
  - American Institute of Research, Whittier, California
  - North Valley Nephrology, Yoba City, California
  - Western Nephrology & Metabolic Bone Disease PC, Arvada, Colorado
  - Western Nephrology & Metabolic Bone Disease PC, Westminister, Colorado
  - Nephrology and Hypertension Associates, Middlebury, Connecticut
  - South Florida Nephrology Group P.A., Coral Springs, Florida
  - Outcomes Research International Inc., Hudson, Florida
  - Nephrology Associates of South Miami, Miami, Florida
  - Nephrology Associates Research Center, Panama City, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Renal Physicians of Georgia PC, Macon, Georgia
  - Boise Kidney & Hypertension Institute, Meridian, Idaho
  - Research by Design LLC, Evergreen Park, Illinois
  - North Suburban Nephrology, Gurnee, Illinois
  - Kansas Nephrology Research Institute LLC, Wichita, Kansas
  - Research Nurse Specialists LLC, Lafayette, Louisiana
  - Lazowski Piotr MD- PC, Plymouth, Massachusetts
  - Fallon Clinic - Winthrop, Worcester, Massachusetts
  - William Beaumont Hospitals, Berkley, Michigan
  - St. Clair Specialty Physicians PC, Detroit, Michigan
  - Nephrology Associates P.C., Columbus, Mississippi
  - Creighton University, Omaha, Nebraska
  - Kantor Nephrology Consultants Ltd., Las Vagas, Nevada
  - Brookdale Physicians Dialysis Associates, Brooklyn, New York
  - Hypertension and Renal Research Group, Buffalo, New York
  - Lower Manhattan Dialysis Center, New York, New York
  - Long Island Hypertension and Nephrology PLLC, Port Washington, New York
  - Wake Nephrology Associates PA, Raleigh, North Carolina
  - University of Cincinnati Medical Center, Cinncinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Humility of Mary Health Partners, Youngstown, Ohio
  - Hypertension and Kidney Specialists, Lancaster, Pennsylvania
  - SC Nephrology & Hypertension Center Inc., Orangeburg, South Carolina
  - Nephrology Associates, Chattanooga, Tennessee
  - Nephrology Associates, Nashville, Tennessee
  - U.S. Renal Care, Arlington, Texas
  - U.S. Renal Care, Burleson, Texas
  - U.S. Renal Care, Fort Worth, Texas
  - Texas Renal Care, Greenville, Texas
  - Ralph Plaza Nephrology, Houston, Texas
  - Dallas Nephrology Associates, Irving, Texas
  - US Renal Care, Mansfield, Texas
  - U.S. Renal Care, McAllen, Texas
  - Dukes Carl, San Antonio, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital and Clinic, Temple, Texas
  - Nephrology Associates of Northern Virginia, Fairfax, Virginia
  - Internal Medicine Kidney and Hypertension Center, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Tidewater Kidney Specialists, Virginia Beach, Virginia
  - Northwest Kidney Center, Seattle, Washington
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Hervey Bay Hospital, Pialba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Royal Melbourne Hospital, Parkville, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Brazil (4):
  - Hospital Universitario da Univ Federal de Juiz de Fora, Juiz de Fora, Minas Gerais
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro, Rio de Janeiro
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo, São Paulo
  - Faculdade de Ciencias Medicas de Sorocaba - Hosp Santa Lucin, Sorocaba, São Paulo
- Canada (9):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Capital District Health Authority, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton, Ontario
  - Clinical Research Solutions Inc., Kitchener, Ontario
  - London Health Science Centre - University Campus Site, London, Ontario
  - St. Michael's Health Care Centre, Toronto, Ontario
  - Exsequi Recherche Clinique, Gatineau, Quebec
  - Hospital Charles LeMoyne, Greenfield Park, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
- France (2):
  - Clinique Mutualiste des Eaux Claires, Grenoble, 38
  - Centre Hospitalier Sud, Amiens, 80
- Germany (6):
  - Gemeinschaftspraxis, Aschaffenburg, Bavaria
  - Klinikum Coburg, Coburg, Bavaria
  - Dialysezentrum Barmbek, Hamburg, Hamburg
  - Dialysepraxis Altona, Hamburg, Hamburg
  - Prager Gerhard, Bad König, Hesse
  - Westpfalz-Klinikum GmbH, Kaiserslautern, Rhineland-Palatinate
- Malta (3):
  - Mater Dei Hospital Medical Outpatient, Birkirkara
  - Mater Dei Hospital Renal Unit, Birkirkara
  - Gozo General Hospital, Gozo
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Wellington Hospital, Wellington
- Poland (5):
  - Szpital Specjalistyczny, Dąbrowa Górnicza
  - NZOZ Avitum-Stacja Dializ Sp.z.o.o, Golub-Dobrzyń
  - NZOZ Miedzynarodowe Centrum Dializ Poznan Odz. Rawicz, Rawicz
  - Euromedic NZOZ Miedzynarodowe, Wroclaw
  - NZOZ Miedzynarodowe Centrum Dializ, Wroclaw
- South Africa (4):
  - Netcare Private Hospital, Bloemfontein, Free State
  - Chris Hani Baragwanath Hospital, Johannesburg, Gauteng
  - St. Augustines Hospital, Durban, KZ-Natal
  - Entabeni Hospital, Durbanville, KZ-Natal
- Spain (2):
  - H Clinic i Provincial, Barcelona
  - HU de Bellvitge, Barcelona